CLINICAL TRIAL: NCT05212909
Title: Anxiety Level Assessment of Anesthesia Providers During COVID-19 Pandemic
Status: Completed | Type: Observational
Sponsor: Augusta University (Other)
Responsible Party: Sponsor
Other Study IDs: 1601067
Record Dates: First submitted 2022-01-25; First posted 2022-01-28 (Actual); Last update posted 2022-02-23 (Actual); Status verified 2022-02

CONDITIONS: Anxiety
Keywords: Anxiety; Mental health; COVID-19; Coronavirus
MeSH Terms: conditions — Anxiety Disorders; Psychological Well-Being; COVID-19; Coronavirus Infections

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: General Anxiety Disorder-7 scale — The General Anxiety Disorder-7 scale was used to evaluate the level of anxiety in anesthesiology providers.

SUMMARY:
Healthcare providers caring for acutely ill or critical patients are exposed to constant stressful situations that can lead to psychiatric manifestations. Depression and anxiety derived from stressful work environments can negatively impact the ability to perform at full capacity directly affecting the quality of care the patients receive.

The Severe Acute Respiratory Syndrome Coronavirus 2 infection created a sudden and deep crisis involving every sector worldwide not only affecting sick patients and the healthcare system but also the economy, politics, food, and drugs and social interactions.

Hospital workers have experienced the crisis first-hand and have witnessed constant death, a decrease in personal protective equipment supplies, exposure to contracting the virus, risk of contagion to others, and overburdened hospital capacity.

The aim of this study is to evaluate how the coronavirus disease 2019 (COVID-19) pandemic has affected healthcare workers. Specifically, to evaluate levels of anxiety and identify factors contributing to anxiety on faculty, residents, and nurse anesthetists in our institution.

DETAILED DESCRIPTION:
The coronavirus disease 2019 (COVID-19) pandemic has affected multiple aspects of everyday life worldwide. Pandemics unleash a societal sense of fear and anxiety. Hence, the COVID-19 pandemic have had a profound impact on mental health. This has led to substantial research on this topic; however, literature evaluating the mental health effects of the pandemic on small groups of people is scarce. Healthcare workers have undergone significant psychological pressure and stress during viral surges of this pandemic. Furthermore, the levels of anxiety vary as the number of cases varies between regions and across time.

After approval by the Institutional Review Board (Protocol # 160167), a cross-sectional study was conducted to identify anxiety levels during the COVID-19 pandemic among anesthesia providers at our institution. The participants included Faculty anesthesiologists, anesthesiology residents, Certified Registered Nurse Anesthetists, and Nurse Anesthetists students. Data were collected from August 26 to September 15, 2020. A questionnaire containing the General Anxiety Disorder-7 (GAD-7) scale, followed by a set of questions with binary answers to evaluate the presence or absence of anxiety-related factors during the COVID-19 pandemic, was administered through direct approach and voluntary participation of the subjects.

ELIGIBILITY:
Inclusion Criteria:

* Anesthesiology providers at Augusta University Medical Center (AU) (Active resident enrolled in the Anesthesiology residency program of Augusta University, Anesthesiologist and Certified Registered Nurse Anesthetist)
* Willingness to participate in the study

Exclusion Criteria:

* Refuses to participate

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Anesthesiology providers at Augusta University Medical Center
Sampling Method: Non-Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
The anxiety levels on anesthesia providers measured by the General Anxiety Disorder 7 scale during COVID-19 pandemic. | one month
  General Anxiety Disorder 7 scale was used to measure anxiety levels.

SECONDARY OUTCOMES:
The association between specific factors such as level of training, occupation, age and gender and the presence of anxiety. | one month
  Specific factors and the association with the presence of anxiety was evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Efrain Riveros-Perez, MD. MBA., Principal Investigator — Augusta University
Locations (1):
- Augusta University Medical Center, Augusta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No